CLINICAL TRIAL: NCT00085111
Title: A Phase I Study of Bevacizumab in Refractory Solid Tumors
Brief Title: Bevacizumab in Treating Young Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01813; ADVL0314; COG-ADVL0314; CDR0000367299; NCI-04-C-0148; U01CA097452 (NIH); NCT00080561 (obsolete NCT alias)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bevacizumab

ARMS (1):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase I trial is studying the side effects and best dose of bevacizumab in treating young patients with refractory solid tumors. Monoclonal antibodies, such as bevacizumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerable dose (MTD) of bevacizumab by dose escalation to a maximum of 15mg/kg, even if MTD is not reached, administered as an intravenous infusion, every 2 weeks to children with refractory solid tumors.

II. To determine the dose-limiting toxicities (DLT) and other toxicities of bevacizumab given on this schedule.

III. To characterize the pharmacokinetic behavior of bevacizumab in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of bevacizumab within the confines of a phase I study.

II. To assess the biologic activity of bevacizumab by measuring levels of total serum VEGF, and parallel angiogenic markers V-CAM-1, ICAM-1, bFGF, and TSP-1 at baseline and at time points post therapy.

III. To explore the biologic effect of bevacizumab on circulating endothelial cells (CECs) and circulating endothelial cell precursors (CECPs).

IV. To determine in archival tumor tissue the expression of VEGF by immunohistochemistry and/or real time PCR.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor at original diagnosis
* Measurable or evaluable* disease
* No known curative therapy exists
* No lymphomas or primary CNS tumors
* No history or clinical evidence of CNS metastasis by head CT scan
* Performance status - Karnofsky 50-100% (patients > 10 years of age)
* Performance status - Lansky 50-100% (patients ≤ 10 years of age)
* At least 8 weeks
* Patients without bone marrow involvement:

  * Absolute neutrophil count ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3 (transfusion independent)
  * Hemoglobin ≥ 8.0 g/dL (RBC transfusion allowed)
* Patients with bone marrow metastases:

  * Platelet count ≥ 75,000/mm^3 (transfusion independent)
  * Granulocytopenia, anemia, and/or mild thrombocytopenia allowed
* No known bleeding diathesis or coagulopathy
* No known thrombophilic condition (e.g., protein S, protein C, or antithrombin III deficiency, Factor V Leiden, Factor II G20210A mutation, homocystinemia, or antiphospholipid antibody syndrome)
* PT or PTT ≤ 1.2 times upper limit of normal (ULN)
* ALT ≤ 5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine clearance or radioisotope glomerular filtrationrate ≥ 70 mL/min
* Creatinine based on age as follows:

  * Creatinine ≤ 0.8 mg/dL (patients ≤ 5 years of age)
  * Creatinine ≤ 1.0 mg/dL (patients 6 to 10 years of age)
  * Creatinine ≤ 1.2 mg/dL (patients 11 to 15 years of age)
  * Creatinine ≤ 1.5 mg/dL (patients > 15 years of age)
* No proteinuria
* 24-hour urine protein ≤ 500 mg
* No history of stroke
* No deep venous or arterial thrombosis within the past 3 months
* No uncontrolled hypertension

  * Hypertension must be well-controlled with stable doses of medication for at least 2 weeks
* No history of myocardial infarction
* No severe or unstable angina
* No transient ischemic attack within the past 6 months
* No cerebrovascular accident within the past 6 months
* No other arterial thromboembolic event within the past 6 months
* No clinically significant or severe peripheral vascular disease
* No pulmonary embolism within the past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* No chronic non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No uncontrolled seizures
* No uncontrolled infection
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Recovered from prior immunotherapy
* More than 1 week since prior growth factors
* At least 2 months since prior stem cell transplantation

  * No evidence of active graft-vs-host disease
* At least 8 weeks since prior monoclonal antibody therapy
* At least 7 days since prior antineoplastic biologic agents
* No prior bevacizumab
* No concurrent prophylactic growth factors
* No other concurrent immunotherapy or biologic therapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent chemotherapy
* Recovered from prior radiotherapy
* At least 4 months since prior craniospinal radiotherapy
* At least 4 months since prior radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 2 weeks since prior local palliative small-port radiotherapy
* No concurrent radiotherapy
* More than 28 days since prior major surgery
* At least 7 days since prior minor surgery (for limited purposes of tissue retrieval) and recovered
* At least 24 hours since prior placement of an indwelling IV catheter
* At least 1 week since prior full-dose anticoagulation therapy, including systemic thrombolytic agents, heparin, low-molecular weight heparin, and warfarin

  * Local intralumenal anticoagulants (e.g., heparin or tissue plasminogen activator) allowed to maintain patency of preexisting, permanent, indwelling IV catheters or peripheral IV catheters for blood sampling
* More than 1 week since prior antipyretic and anti-inflammatory medications (except acetaminophen)
* No concurrent full-dose anticoagulation therapy
* No concurrent anti-inflammatory medication
* Concurrent acetaminophen allowed
* No other concurrent cancer therapy
* No other concurrent investigational agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2003-12; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined based on the dose-limiting toxicities graded according to Common Terminology Criteria for Adverse Events v3.0 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bender, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States